CLINICAL TRIAL: NCT06619080
Title: Ecoguided Genicular Nerve Block in Patients With Knee Osteoarthritis by Local Anesthetic or by Combination of Local Anesthetic and Corticoid: Placebo-Controlled Randomized Blind Clinical Trial
Brief Title: Ecoguided Genicular Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Fundación Alcorcón (Other)
Responsible Party: Principal Investigator, Claudia de la Fuente Escudero, Consultant Specialist in Physical Medicine and Rehabilitation, Hospital Universitario Fundación Alcorcón
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22/149; 2022-003885-19 (EudraCT Number)
Record Dates: First submitted 2024-08-30; First posted 2024-10-01 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee/Rehabilitation
Keywords: "Nerve Block"[MeSH Terms]; "Exercise"[MeSH Terms]; Ultrasound-guided infiltration; Genicular nerves
MeSH Terms: conditions — Osteoarthritis | interventions — Bupivacaine; Adrenal Cortex Hormones; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Study Design Type of Study: Pilot randomized controlled experimental clinical trial. Number of Groups: Three parallel treatment arms.
  Intervention Groups:
  Group 1: Block with 0.5% bupivacaine and corticosteroid (triamcinolone). Group 2: Block with 0.5% bupivacaine. Group 3 (Control): Block with saline solution. Randomization
  Technique Description:
  Patient Position: Supine with knee extended. Ultrasound-Guided Localization: Use of ultrasound with Doppler to locate genicular nerves and associated arteries.
  Injection Points:
  Superior medial and lateral genicular nerves: Femoral condyle and junction with the femoral shaft.
  Inferior medial genicular nerve: Medial tibial-femoral joint line.
  Injection Doses:
  Group 1: 2.5 mL of 0.5% bupivacaine + 20 mg of triamcinolone. Group 2: 2.5 mL of 0.5% bupivacaine. Group 3: 2.5 mL of saline solution.
Who Masked: Participant, Investigator
Masking Description: Concealed Random Assignment: Participants will be assigned to one of three treatment groups using a computer-generated sequence. Opaque, sequentially numbered envelopes with treatment assignments will be opened after patient inclusion.
  Blinding of Participants: Participants will not know the specific injection content (bupivacaine with or without corticosteroids, or saline). They will only know they are receiving one of the study interventions.
  Blinding of Investigators: Investigators for initial evaluation and follow-up will not administer treatments. Independent personnel will prepare and administer treatments without evaluating outcomes.
  Blind Evaluations: Pain and functionality (VAS, KOOS, WOMAC, KUJALA) will be assessed by blinded investigators. Follow-up consultations will be handled by personnel unaware of treatment details.
  Documentation and Verification: Secure treatment assignment records will be accessible only to the data and safety monitoring committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Block with 0.5% bupivacaine and corticosteroid (triamcinolone). (Active Comparator): Injection Doses: 2.5 mL of 0.5% bupivacaine + 20 mg of triamcinolone.
  Interventions: Drug: Genicular nerve block with bupivacaine and corticosteroids
- Group 2: Block with 0.5% bupivacaine. (Active Comparator): Injection Doses: 2.5 mL of 0.5% bupivacaine.
  Interventions: Drug: Genicular nerve block with bupivacaine
- Group 3 (Control): Block with saline solution. (Placebo Comparator): Injection Doses: 2.5 mL of saline solution.
  Interventions: Drug: Genicular nerve block with saline

INTERVENTIONS:
Drug: Genicular nerve block with bupivacaine and corticosteroids — - GROUP 1:Genicular Nerve Block with Bupivacaine and Corticosteroids: 2.5 mL at three genicular nerve points.
  All injections are ultrasound-guided and administered once. The primary outcome is pain reduction, measured using NRS, KOOS, WOMAC, and KUJALA scales at 4, 12, and 24 weeks post-injection. Follow-up includes phone and in-person consultations to monitor pain, functionality, and adverse effects.
  Arms: Group 1: Block with 0.5% bupivacaine and corticosteroid (triamcinolone).
Drug: Genicular nerve block with bupivacaine — - GROUP 2: Genicular Nerve Block with Bupivacaine: 2.5 mL at three genicular nerve points.
  All injections are ultrasound-guided and administered once. The primary outcome is pain reduction, measured using NRS, KOOS, WOMAC, and KUJALA scales at 4, 12, and 24 weeks post-injection. Follow-up includes phone and in-person consultations to monitor pain, functionality, and adverse effects.
  Arms: Group 2: Block with 0.5% bupivacaine.
Drug: Genicular nerve block with saline — - GROUP 3: Genicular Nerve Block with Saline: 2.5 mL at three genicular nerve points.
  All injections are ultrasound-guided and administered once. The primary outcome is pain reduction, measured using NRS, KOOS, WOMAC, and KUJALA scales at 4, 12, and 24 weeks post-injection. Follow-up includes phone and in-person consultations to monitor pain, functionality, and adverse effects.
  Arms: Group 3 (Control): Block with saline solution.

SUMMARY:
Osteoarthritis is a pathology with high prevalence in the world and is increasing due to sedentary lifestyles. Recent researches that claim for conservative treatment have shown the utility of genicular nerve blocks for relief of chronic knee pain.

Likewise, the ultrasound-guided technique has been more popular among professionals in recent years due to its low cost and safety.

This pilot study tries to evaluate if the infiltration of local anesthetic could avoid the use of corticosteroids with the secondary effects that they entail, therefore, it is carried out with the intention of estimating the size of the effect and the use of the variable response for later carrying out a clinical trial.

For this, we propose the comparative analysis of three randomized groups of patients (n=90), where all of them will perform a quadriceps strengthening exercise at home. Moreover, we will assess the reduction of pain through the visual analog scale (VAS) after the genicular nerve block with ultrasound-guided infiltration. Group 1 (n=30) will be infiltrated with local anesthetic and steroid, group 2 (n=30) with local anesthetic and group 3 (n=30), as a control group, will receive physiological saline. We will also record demographic data, functionality and mood using validated scales.

DETAILED DESCRIPTION:
Osteoarthritis affects approximately 302 million people worldwide, with the knee, hip, and hands being the most commonly affected areas. Knee osteoarthritis is highly prevalent and increasing in the region due to aging, obesity, and the progressive sedentary lifestyle of the population. According to recent epidemiological studies, it has a prevalence of 29.3% in the Spanish population.

Currently, multiple treatment options are available, ranging from conservative measures to surgical procedures. Within conservative treatment, various tools benefit patients and may even avoid the need for surgery. These non-surgical options include patient education, weight control, physical exercise, orthotics, oral analgesics, topical anti-inflammatories, and interventional procedures. However, there are no prior studies demonstrating the advantages of one over another, and many do not follow up beyond three months.

When conservative treatment is ineffective, surgical intervention is usually considered. Therapeutic options include knee arthroscopy, high tibial osteotomy, total knee replacement, and unicompartmental knee replacement in patients without lateral compartment disease.

Traditionally, rest and caution in exercise were recommended for knee osteoarthritis pain. However, this paradigm has been strongly rejected. One of the current first-line treatments for knee osteoarthritis is physical exercise, with quadriceps strengthening being the most indicated. Most patients seek recommendations on what type of exercise to perform, including the duration, intensity, and frequency for better adherence. No exercise has been shown to be superior to another, with the most studied being yoga and tai chi exercises.

Despite the well-documented benefits of exercise for this condition, one emerging procedure for pain management is the genicular nerve block. This treatment option can facilitate progress in the exercise program. It is also indicated for patients who have previously had successful genicular block, those who do not wish to undergo surgery, those not eligible for surgery, or even post-surgical patients for better pain control.

The term "genicular nerves" refers to a group of nerves responsible for the sensory innervation of the knee joint capsule and the internal and external ligaments. The superior and inferior medial genicular nerves are sensory branches of the tibial nerve, whereas the superior and inferior lateral genicular nerves are branches of the common peroneal nerve. These nerves are named after the arteries they accompany, which are located using ultrasound during the procedure.

Genicular nerve block is a simple technique that significantly reduces opioid consumption in patients undergoing total knee arthroplasty within the first 24 hours. It also provides temporary relief that allows progression in the rehabilitation program through a structured exercise regimen. This technique involves injecting medication into the genicular nerves, locating the genicular artery using Doppler ultrasound. Various cadaveric studies have investigated the anatomical distribution of the descending genicular artery and the nerves accompanying its branches.

Some authors suggest that up to 10 points may need to be blocked for complete coverage. However, this is not feasible in routine clinical practice. Most studies target three sensory nerves of the knee: the superior lateral genicular nerve, the superior medial genicular nerve, and the inferior medial genicular nerve. In most studies, 2 to 3 ml of local anesthetic is administered per point. It has been shown that 0.5 ml of injected fluid spreads within the tissue over an area of 6 cm², likely covering more nerve targets with 2 ml. Typically, the procedure involves infiltrating local anesthetic (lidocaine, bupivacaine, ropivacaine, levobupivacaine) and 20 mg of corticosteroid (triamcinolone).

In this study, bupivacaine is chosen as the local anesthetic, as it inhibits prostaglandin production by binding to the E2 receptor, providing an anti-inflammatory effect. It is a lipophilic amide-type anesthetic with 100% bioavailability and a longer duration than other local anesthetics. Additionally, it produces a more significant blockade of sensory and sympathetic nerve fibers than motor fibers, differentiating it from other local anesthetics.

Recent guidelines for the treatment of knee osteoarthritis highlight the recommendation of intra-articular corticosteroid injections. However, several studies mention that systemic and local corticosteroid effects can cause adverse effects such as skin atrophy, hypertension, insulin resistance, decreased bone mineralization, and septic arthritis, among others. Nonetheless, these effects have not demonstrated a direct relationship with pain, functionality, or radiological changes.

The clinical benefit of corticosteroid administration compared to local anesthesia alone remains unclear. Given the potential adverse effects, corticosteroids may not be suitable as adjuvants. Therefore, genicular nerve block using local anesthetic alone proves to be a promising technique, avoiding the use of corticosteroids and not being an intra-articular procedure.

A study is proposed at a tertiary hospital in the Community of Madrid (Hospital Universitario Fundación Alcorcón). Considering the absence of previous studies that evaluate and quantify the three described treatment options, this study aims to address this objective through a pilot experimental randomized controlled trial. All patients will receive guidelines for an exercise program, and the outcomes of adding genicular nerve block with and without corticosteroid will be assessed. This unprecedented study could identify the optimal treatment for this prevalent and debilitating condition in a significant portion of the population. Additionally, it will help optimize resource allocation for these patients by identifying the best therapeutic target, thus avoiding unnecessary resource consumption

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Anterior knee pain of patellofemoral origin and/or femorotibial compartment osteoarthritis with no previous response to pharmacological treatment (oral and/or topical)
* Pain duration of 3 months
* Pain assessment scale (Numerical Rating Scale) ≥ 5
* Radiological study with Kellgren-Lawrence classification > 2

Exclusion Criteria:

* Allergy to the active ingredients and excipients of: bupivacaine, triamcinolone, or saline solution
* Patients who have undergone total or unicompartmental knee replacement surgery
* Viscosupplementation or intra-articular corticosteroid injection within the last 3 months
* Pregnant women or those suspected of being pregnant
* Cognitive impairment or additional neuropsychiatric symptoms
* Failure to sign informed consent or revocation of it
* Patients with heart disease requiring blockade with levobupivacaine
* Inability to write, speak, or read in Spanish
* Active tumoral or infectious pathology
* Osteoarthritis secondary to inflammatory pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Reduction in Pain | Baseline, 4 weeks, 12 weeks, and 24 weeks post-procedure
  * Measurement Tool: Numeric Rating Scale (NRS)
  * Minimum Value: 0
  * Maximum Value: 10
  * Interpretation: Higher scores indicate worse pain.

SECONDARY OUTCOMES:
Mood Evaluation | Baseline, 4 weeks, 12 weeks, and 24 weeks post-procedure
  EVEA (Emotional State Evaluation Scale) [Time Frame: Baseline, 4 weeks, 12 weeks, and 24 weeks post-procedure]
  * Minimum Value: 0
  * Maximum Value: 100
  * Interpretation: Higher scores indicate a worse emotional state
Physical Examination | Baseline, 4 weeks, 12 weeks, and 24 weeks post-procedure
  Degrees of Knee Flexion and Extension [Time Frame: Baseline, 4 weeks, 12 weeks, and 24 weeks post-procedure]
  * Measurement Tool: Goniometer
  * Minimum Value: 0 degrees (full extension)
  * Maximum Value: 140 degrees (full flexion)
  * Interpretation: Higher values indicate greater knee flexion. Description: Physical examination to assess changes in the range of motion of the knee
Functionality Improvement | Baseline, 4 weeks, 12 weeks, and 24 weeks post-procedure
  - KOOS (Knee Injury and Osteoarthritis Outcome Score) [Time Frame: Baseline, 4 weeks, 12 weeks, and 24 weeks post-procedure]
  * Minimum Value: 0
  * Maximum Value: 100
  * Interpretation: Higher scores indicate better knee function.
Functionality improvement | Baseline, 4 weeks, 12 weeks, and 24 weeks post-procedure
  - WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index Score)
  * Minimum Value: 0
  * Maximum Value: 96
  * Interpretation: Lower scores indicate better knee function.
Functionality Improvement | Baseline, 4 weeks, 12 weeks, and 24 weeks post-procedure
  KUJALA Scale:
  * Minimum Value: 0
  * Maximum Value: 100
  * Interpretation: Higher scores indicate better knee function
Incidence of Adverse Events | Through study completion, an average of 1 year
  Monitoring and documentation of any adverse events to evaluate the safety of the interventions.
Demographic and clinical variables | Baseline
  2. Sex [Time Frame: Baseline]
  o Measurement: Gender (Male/Female)
Demographic and Clinical Variables | Baseline
  1. Age [Time Frame: Baseline]
  o Measurement: Age in years
Demographic and clinical variables | Baseline
  3. Hypertension [Time Frame: Baseline]
  o Measurement: Presence of hypertension (Yes/No)
Demographic and clinical variables | Baseline
  Diabetes Mellitus [Time Frame: Baseline]
  o Measurement: Presence of diabetes mellitus (Yes/No)
Demographic and clinical variables | Baseline
  Body Mass Index (BMI) [Time Frame: Baseline]
  * Measurement: BMI in kg/m²
  * Minimum Value: Variable
  * Maximum Value: Variable
  * Interpretation: Higher values indicate higher body weight relative to height.
Demographic and clinical variables | Baseline
  Anticoagulation Status [Time Frame: Baseline]
  o Measurement: Use of anticoagulants (Yes/No)
Demographic and clinical variables | Baseline
  Laterality (Left or Right Knee) [Time Frame: Baseline]
  o Measurement: Knee affected (Left/Right)
Demographic and clinical variables | Baseline
  Duration of Symptoms [Time Frame: Baseline]
  o Measurement: Duration of knee pain in months
Demographic and clinical variables | Baseline
  Previous Intra-Articular Injections [Time Frame: Baseline]
  o Measurement: History of previous injections (Yes/No)
Analgesic Medication Use | Through study completion, an average of 1 year
  Description: Analysis of the reduction in the use of analgesic medications post-procedure
Demographic and clinical variables | Baseline
  10. Use of Assistive Walking Devices Measurement: Yes/No
Analgesic Medication Use | Through study completion, an average of 1 year
  o Measurement: Type of analgesic medication consumed

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Plan Description: Individual participant data (IPD) collected in this study will not be shared. The reasons for this decision include:
  * Privacy Concerns: Protecting participant confidentiality is paramount. Sharing IPD could potentially compromise participant privacy
  * Proprietary Information: The data collected includes proprietary information that cannot be disclosed due to legal or contractual reasons
  * Data Quality and Integrity: To maintain the accuracy and integrity of the data, sharing IPD might lead to misuse or misinterpretation
  * Institutional Policies: Institutional policies restrict the sharing of data to comply with ethical and regulatory standards
  * Resource Limitations: The study team lacks the resources to manage and facilitate IPD sharing effectively
  Access Criteria: As IPD will not be shared, there are no access criteria.

REFERENCES:
- [Background] Luan L, El-Ansary D, Adams R, Wu S, Han J. Knee osteoarthritis pain and stretching exercises: a systematic review and meta-analysis. Physiotherapy. 2022 Mar;114:16-29. doi: 10.1016/j.physio.2021.10.001. Epub 2021 Oct 11. PMID 35091326
- [Background] Marriott KA, Hall M, Maciukiewicz JM, Almaw RD, Wiebenga EG, Ivanochko NK, Rinaldi D, Tung EV, Bennell KL, Maly MR. Are the Effects of Resistance Exercise on Pain and Function in Knee and Hip Osteoarthritis Dependent on Exercise Volume, Duration, and Adherence? A Systematic Review and Meta-Analysis. Arthritis Care Res (Hoboken). 2024 Jun;76(6):821-830. doi: 10.1002/acr.25313. Epub 2024 Apr 15. PMID 38317328
- [Background] Messier SP, Mihalko SL, Beavers DP, Nicklas BJ, DeVita P, Carr JJ, Hunter DJ, Lyles M, Guermazi A, Bennell KL, Loeser RF. Effect of High-Intensity Strength Training on Knee Pain and Knee Joint Compressive Forces Among Adults With Knee Osteoarthritis: The START Randomized Clinical Trial. JAMA. 2021 Feb 16;325(7):646-657. doi: 10.1001/jama.2021.0411. PMID 33591346
- [Background] Mo L, Jiang B, Mei T, Zhou D. Exercise Therapy for Knee Osteoarthritis: A Systematic Review and Network Meta-analysis. Orthop J Sports Med. 2023 Jun 5;11(5):23259671231172773. doi: 10.1177/23259671231172773. eCollection 2023 May. PMID 37346776
- [Background] Patterson BE, Girdwood MA, West TJ, Bruder AM, Oiestad BE, Juhl C, Culvenor AG. Muscle strength and osteoarthritis of the knee: a systematic review and meta-analysis of longitudinal studies. Skeletal Radiol. 2023 Nov;52(11):2085-2097. doi: 10.1007/s00256-022-04266-4. Epub 2022 Dec 23. PMID 36562820
- [Background] Puts S, Liberman K, Leysen L, Forti L, Muyldermans E, Vaes P, Nijs J, Beckwee D, Bautmans I. Exercise-induced effects on inflammatory markers and brain-derived neurotrophic factor in patients with knee osteoarthritis. A systematic review with meta-analysis. Exerc Immunol Rev. 2023;29:22-53. PMID 37358362
- [Background] Raposo F, Ramos M, Lucia Cruz A. Effects of exercise on knee osteoarthritis: A systematic review. Musculoskeletal Care. 2021 Dec;19(4):399-435. doi: 10.1002/msc.1538. Epub 2021 Mar 5. PMID 33666347
- [Background] Reichenbach S, Juni P, Hincapie CA, Schneider C, Meli DN, Schurch R, Streit S, Lucas C, Mebes C, Rutjes AWS, da Costa BR. Effect of transcutaneous electrical nerve stimulation (TENS) on knee pain and physical function in patients with symptomatic knee osteoarthritis: the ETRELKA randomized clinical trial. Osteoarthritis Cartilage. 2022 Mar;30(3):426-435. doi: 10.1016/j.joca.2021.10.015. Epub 2021 Nov 23. PMID 34826572
- [Background] Rezasoltani Z, Azizi S, Najafi S, Sanati E, Dadarkhah A, Abdorrazaghi F. Physical therapy, intra-articular dextrose prolotherapy, botulinum neurotoxin, and hyaluronic acid for knee osteoarthritis: randomized clinical trial. Int J Rehabil Res. 2020 Sep;43(3):219-227. doi: 10.1097/MRR.0000000000000411. PMID 32776763
- [Background] Rocha TC, Ramos PDS, Dias AG, Martins EA. The Effects of Physical Exercise on Pain Management in Patients with Knee Osteoarthritis: A Systematic Review with Metanalysis. Rev Bras Ortop (Sao Paulo). 2020 Oct;55(5):509-517. doi: 10.1055/s-0039-1696681. Epub 2019 Sep 23. PMID 33093712
- [Background] Santos ACG, Caiado VDS, Moreira-Marconi E, Teixeira-Silva Y, De Meirelles AG, Seixas A, Lacerda ACR, Sonza A, Mendonca VA, Bernardo-Filho M, De Sa-Caputo DDC. The Influence of Physical Exercises on the Flexibility of Older Individuals with Knee Osteoarthritis: A Systematic Review. Iran J Public Health. 2024 Feb;53(2):255-267. doi: 10.18502/ijph.v53i2.14911. PMID 38894836
- [Background] Si J, Sun L, Li Z, Zhu W, Yin W, Peng L. Effectiveness of home-based exercise interventions on pain, physical function and quality of life in individuals with knee osteoarthritis: a systematic review and meta-analysis. J Orthop Surg Res. 2023 Jul 17;18(1):503. doi: 10.1186/s13018-023-04004-z. PMID 37461112
- [Background] Sinatti P, Sanchez Romero EA, Martinez-Pozas O, Villafane JH. Effects of Patient Education on Pain and Function and Its Impact on Conservative Treatment in Elderly Patients with Pain Related to Hip and Knee Osteoarthritis: A Systematic Review. Int J Environ Res Public Health. 2022 May 19;19(10):6194. doi: 10.3390/ijerph19106194. PMID 35627729
- [Background] Smith KM, Massey BJ, Young JL, Rhon DI. What are the unsupervised exercise adherence rates in clinical trials for knee osteoarthritis? A systematic review. Braz J Phys Ther. 2023 Jul-Aug;27(4):100533. doi: 10.1016/j.bjpt.2023.100533. Epub 2023 Aug 12. PMID 37597491
- [Background] Weng Q, Goh SL, Wu J, Persson MSM, Wei J, Sarmanova A, Li X, Hall M, Doherty M, Jiang T, Zeng C, Lei G, Zhang W. Comparative efficacy of exercise therapy and oral non-steroidal anti-inflammatory drugs and paracetamol for knee or hip osteoarthritis: a network meta-analysis of randomised controlled trials. Br J Sports Med. 2023 Aug;57(15):990-996. doi: 10.1136/bjsports-2022-105898. Epub 2023 Jan 2. PMID 36593092
- [Background] Wolf DF, Carvalho C, Moreira Padovez RFC, Braz de Oliveira MP, Mendes da Silva Serrao PR. Effects of physical exercise on muscle function of the knee, pain and quality of life in postmenopausal women with knee osteoarthritis: A systematic review with meta-analysis. Musculoskelet Sci Pract. 2024 Jun;71:102929. doi: 10.1016/j.msksp.2024.102929. Epub 2024 Mar 11. PMID 38489855
- [Background] Zhang L, Wang Y, Ye T, Hu Y, Wang S, Qian T, Wu C, Yue S, Sun X, Zhang Y. Quality of clinical practice guidelines relevant to rehabilitation of knee osteoarthritis: A systematic review. Clin Rehabil. 2023 Jul;37(7):986-1008. doi: 10.1177/02692155221144892. Epub 2022 Dec 20. PMID 36540949
- [Background] Zhang ZY, Huang L, Tian L, Yi J, Gao M, Wang XQ, Jiang JJ, Liu ZL. Home-based vs center-based exercise on patient-reported and performance-based outcomes for knee osteoarthritis: a systematic review with meta-analysis. Front Public Health. 2024 Mar 14;12:1360824. doi: 10.3389/fpubh.2024.1360824. eCollection 2024. PMID 38550325
- [Background] Zhu GC, Chen KM, Belcastro F. Comparing Different Stretching Exercises on Pain, Stiffness, and Physical Function Disability in Older Adults With Knee Osteoarthritis. Arch Phys Med Rehabil. 2024 May;105(5):953-962. doi: 10.1016/j.apmr.2023.07.001. Epub 2023 Jul 17. PMID 37467937
- [Background] Tan B, Yan Y, Zhou Q, Ran Q, Chen H, Sun S, Lu W, Chen W, Wang J. Kinesitherapy for Knee Osteoarthritis Patients Physical and Psychological Health Based on "Traditional Chinese Exercise" Management Modalities: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Orthop Surg. 2024 Jan;16(1):3-16. doi: 10.1111/os.13920. Epub 2023 Nov 29. PMID 38018392
- [Background] Tayfur B, Charuphongsa C, Morrissey D, Miller SC. Neuromuscular joint function in knee osteoarthritis: A systematic review and meta-analysis. Ann Phys Rehabil Med. 2023 Mar;66(2):101662. doi: 10.1016/j.rehab.2022.101662. Epub 2022 Dec 1. PMID 35364316
- [Background] Thomas DT, R S, Prabhakar AJ, Dineshbhai PV, Eapen C. Hip abductor strengthening in patients diagnosed with knee osteoarthritis - a systematic review and meta-analysis. BMC Musculoskelet Disord. 2022 Jun 29;23(1):622. doi: 10.1186/s12891-022-05557-6. PMID 35768802
- [Background] Thorlund JB, Simic M, Pihl K, Berthelsen DB, Day R, Koes B, Juhl CB. Similar Effects of Exercise Therapy, Nonsteroidal Anti-inflammatory Drugs, and Opioids for Knee Osteoarthritis Pain: A Systematic Review with Network Meta-analysis. J Orthop Sports Phys Ther. 2022 Apr;52(4):207-216. doi: 10.2519/jospt.2022.10490. PMID 35442752
- [Background] Torstensen TA, Osteras H, LoMartire R, Rugelbak GM, Grooten WJA, Ang BO. High- Versus Low-Dose Exercise Therapy for Knee Osteoarthritis : A Randomized Controlled Multicenter Trial. Ann Intern Med. 2023 Feb;176(2):154-165. doi: 10.7326/M22-2348. Epub 2023 Jan 24. PMID 36689746
- [Background] Vassao PG, Parisi J, Penha TFC, Balao AB, Renno ACM, Avila MA. Association of photobiomodulation therapy (PBMT) and exercises programs in pain and functional capacity of patients with knee osteoarthritis (KOA): a systematic review of randomized trials. Lasers Med Sci. 2021 Sep;36(7):1341-1353. doi: 10.1007/s10103-020-03223-8. Epub 2021 Jan 3. PMID 33392780
- [Background] Henriksen M, Nielsen SM, Christensen R, Kristensen LE, Bliddal H, Bartholdy C, Boesen M, Ellegaard K, Hunter DJ, Altman R, Bandak E. Who are likely to benefit from the Good Life with osteoArthritis in Denmark (GLAD) exercise and education program? An effect modifier analysis of a randomised controlled trial. Osteoarthritis Cartilage. 2023 Jan;31(1):106-114. doi: 10.1016/j.joca.2022.09.001. Epub 2022 Sep 8. PMID 36089229
- [Background] Henriksen M, Christensen R, Kristensen LE, Bliddal H, Bartholdy C, Boesen M, Ellegaard K, Guldberg-Moller J, Hunter DJ, Altman R, Bandak E. Exercise and education vs intra-articular saline for knee osteoarthritis: a 1-year follow-up of a randomized trial. Osteoarthritis Cartilage. 2023 May;31(5):627-635. doi: 10.1016/j.joca.2022.12.011. Epub 2023 Jan 16. PMID 36657659
- [Background] Hall M, Dobson F, Van Ginckel A, Nelligan RK, Collins NJ, Smith MD, Ross MH, Smits E, Bennell KL. Comparative effectiveness of exercise programs for psychological well-being in knee osteoarthritis: A systematic review and network meta-analysis. Semin Arthritis Rheum. 2021 Oct;51(5):1023-1032. doi: 10.1016/j.semarthrit.2021.07.007. Epub 2021 Jul 26. PMID 34416624
- [Background] Guede-Rojas F, Benavides-Villanueva A, Salgado-Gonzalez S, Mendoza C, Arias-Alvarez G, Soto-Martinez A, Carvajal-Parodi C. Effect of strength training on knee proprioception in patients with knee osteoarthritis: A systematic review and meta-analysis. Sports Med Health Sci. 2023 Nov 7;6(2):101-110. doi: 10.1016/j.smhs.2023.10.005. eCollection 2024 Jun. PMID 38708322
- [Background] Donec V, Kubilius R. The effectiveness of Kinesio Taping(R) for mobility and functioning improvement in knee osteoarthritis: a randomized, double-blind, controlled trial. Clin Rehabil. 2020 Jul;34(7):877-889. doi: 10.1177/0269215520916859. Epub 2020 May 6. PMID 32372651
- [Background] Denham-Jones L, Gaskell L, Spence N, Pigott T. A systematic review of the effectiveness of Pilates on pain, disability, physical function, and quality of life in older adults with chronic musculoskeletal conditions. Musculoskeletal Care. 2022 Mar;20(1):10-30. doi: 10.1002/msc.1563. Epub 2021 May 24. PMID 34028164
- [Background] de Zwart AH, Dekker J, Roorda LD, van der Esch M, Lips P, van Schoor NM, Heijboer AC, Turkstra F, Gerritsen M, Hakkinen A, Bennell K, Steultjens MP, Lems WF, van der Leeden M. High-intensity versus low-intensity resistance training in patients with knee osteoarthritis: A randomized controlled trial. Clin Rehabil. 2022 Jul;36(7):952-967. doi: 10.1177/02692155211073039. Epub 2022 Mar 25. PMID 35331018
- [Background] Ceballos-Laita L, Lahuerta-Martin S, Carrasco-Uribarren A, Cabanillas-Barea S, Hernandez-Lazaro H, Perez-Guillen S, Jimenez-Del-Barrio S. Strength Training vs. Aerobic Training for Managing Pain and Physical Function in Patients with Knee Osteoarthritis: A Systematic Review and Meta-Analysis. Healthcare (Basel). 2023 Dec 22;12(1):33. doi: 10.3390/healthcare12010033. PMID 38200939
- [Background] Carvalho MTX, Guesser Pinheiro VH, Alberton CL. Effectiveness of neuromuscular electrical stimulation training combined with exercise on patient-reported outcomes measures in people with knee osteoarthritis: A systematic review and meta-analysis. Physiother Res Int. 2024 Jan;29(1):e2062. doi: 10.1002/pri.2062. Epub 2023 Nov 5. PMID 37926438
- [Background] Bennell KL, Nelligan RK, Kimp AJ, Schwartz S, Kasza J, Wrigley TV, Metcalf B, Hodges PW, Hinman RS. What type of exercise is most effective for people with knee osteoarthritis and co-morbid obesity?: The TARGET randomized controlled trial. Osteoarthritis Cartilage. 2020 Jun;28(6):755-765. doi: 10.1016/j.joca.2020.02.838. Epub 2020 Mar 19. PMID 32200051
- [Background] Misseri G, Gregoretti C, Lo Bianco G. Review of Evaluation and Treatment of Knee Pain. JAMA. 2024 Feb 27;331(8):706-707. doi: 10.1001/jama.2023.27754. No abstract available. PMID 38411652
- [Background] Bandak E, Christensen R, Overgaard A, Kristensen LE, Ellegaard K, Guldberg-Moller J, Bartholdy C, Hunter DJ, Altman R, Bliddal H, Henriksen M. Exercise and education versus saline injections for knee osteoarthritis: a randomised controlled equivalence trial. Ann Rheum Dis. 2022 Apr;81(4):537-543. doi: 10.1136/annrheumdis-2021-221129. Epub 2021 Nov 29. PMID 34844929
- [Background] Rambhia M, Chen A, Kumar AH, Bullock WM, Bolognesi M, Gadsden J. Ultrasound-guided genicular nerve blocks following total knee arthroplasty: a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2021 Oct;46(10):862-866. doi: 10.1136/rapm-2021-102667. Epub 2021 Jul 14. PMID 34261807
- [Background] Sebastian MP, Dsouza SL, Aranburu Uriarte O. IPACK and genicular nerves block: which nerves are we targeting? Reg Anesth Pain Med. 2022 Mar;47(3):201-202. doi: 10.1136/rapm-2021-103105. Epub 2021 Sep 13. No abstract available. PMID 34518371
- [Background] Fletcher A, Moore KJ, Stensby JD, Hulbert A, Saemi AM, Davis RM, Bhat AP. The Pain Crisis: Interventional Radiology's Role in Pain Management. AJR Am J Roentgenol. 2021 Sep;217(3):676-690. doi: 10.2214/AJR.20.24265. Epub 2020 Sep 23. PMID 32966117
- [Background] Fonkoue L, Behets C, Steyaert A, Kouassi JK, Detrembleur C, Cornu O. Anatomical study of the descending genicular artery and implications for image-guided interventions for knee pain. Clin Anat. 2021 May;34(4):634-643. doi: 10.1002/ca.23680. Epub 2020 Sep 21. PMID 32920906
- [Background] Fitzpatrick B, Cowling M, Poliak-Tunis M, Miller K. Effect of Genicular Nerve Radiofrequency Ablation for Knee Osteoarthritis: A Retrospective Chart Review. WMJ. 2021 Jul;120(2):156-159. PMID 34255959
- [Background] Kim PY, Cohen SP. Genicular Nerve Blocks and Radiofrequency Ablation for Knee Osteoarthritis: More Nerves, More Questions. Pain Med. 2021 May 21;22(5):1019-1021. doi: 10.1093/pm/pnab022. No abstract available. PMID 33538816
- [Background] Cankurtaran D, Karaahmet OZ, Yildiz SY, Eksioglu E, Dulgeroglu D, Unlu E. Comparing the effectiveness of ultrasound guided versus blind genicular nerve block on pain, muscle strength with isokinetic device, physical function and quality of life in chronic knee osteoarthritis: a prospective randomized controlled study. Korean J Pain. 2020 Jul 1;33(3):258-266. doi: 10.3344/kjp.2020.33.3.258. PMID 32606270
- [Background] Ferreira-Dos-Santos G, Hurdle MB, Gupta S, Tran J, Agur AMR, Clendenen SR. Revisiting the Genicular Nerve Block: An Up-to-Date Guide Utilizing Ultrasound Guidance and Peripheral Nerve Stimulation - Anatomy Description and Technique Standardization. Pain Physician. 2021 Mar;24(2):E177-E183. PMID 33740351
- [Background] Shanahan EM, Robinson L, Lyne S, Woodman R, Cai F, Dissanayake K, Paddick K, Cheung G, Voyvodic F. Genicular Nerve Block for Pain Management in Patients With Knee Osteoarthritis: A Randomized Placebo-Controlled Trial. Arthritis Rheumatol. 2023 Feb;75(2):201-209. doi: 10.1002/art.42384. Epub 2022 Nov 11. PMID 36369781
- [Background] Zaragoza G, Solorzano-Flores SY, Pineda C, Soto-Fajardo C. Ultrasound-guided genicular nerve block a new treatment in rheumatology for knee osteoarthritis pain. Rheumatol Int. 2022 Sep;42(9):1663-1664. doi: 10.1007/s00296-022-05162-9. Epub 2022 Jun 17. No abstract available. PMID 35713678
- [Background] Yilmaz V, Umay E, Gundogdu I, Aras B. The comparison of efficacy of single intraarticular steroid injection versus the combination of genicular nerve block and intraarticular steroid injection in patients with knee osteoarthritis: a randomised study. Musculoskelet Surg. 2021 Apr;105(1):89-96. doi: 10.1007/s12306-019-00633-y. Epub 2019 Dec 11. PMID 31828590
- [Background] DemIr Y, Guzelkucuk U, Tezel K, AydemIr K, Taskaynatan MA. A Different Approach to the Management of Osteoarthritis in the Knee: Ultrasound Guided Genicular Nerve Block. Pain Med. 2017 Jan 1;18(1):181-183. doi: 10.1093/pm/pnw177. No abstract available. PMID 27492742
- [Background] Qudsi-Sinclair S, Borras-Rubio E, Abellan-Guillen JF, Padilla Del Rey ML, Ruiz-Merino G. A Comparison of Genicular Nerve Treatment Using Either Radiofrequency or Analgesic Block with Corticosteroid for Pain after a Total Knee Arthroplasty: A Double-Blind, Randomized Clinical Study. Pain Pract. 2017 Jun;17(5):578-588. doi: 10.1111/papr.12481. Epub 2016 Sep 19. PMID 27641918
- [Background] Pietrantoni P, Cunat T, Nuevo-Gayoso M, Martin N, Tio M, Basora M, Sastre S, Sala-Blanch X. Ultrasound-guided genicular nerves block: an analgesic alternative to local infiltration analgesia for total knee arthroplasty: A noninferiority, matched cohort study. Eur J Anaesthesiol. 2021 Aug 1;38(Suppl 2):S130-S137. doi: 10.1097/EJA.0000000000001546. PMID 34038916
- [Background] Kidd VD, Strum SR, Strum DS, Shah J. Genicular Nerve Radiofrequency Ablation for Painful Knee Arthritis: The Why and the How. JBJS Essent Surg Tech. 2019 Mar 13;9(1):e10. doi: 10.2106/JBJS.ST.18.00016. eCollection 2019 Mar 26. PMID 31333900
- [Background] Husted RS, Troelsen A, Husted H, Gronfeldt BM, Thorborg K, Kallemose T, Rathleff MS, Bandholm T. Knee-extensor strength, symptoms, and need for surgery after two, four, or six exercise sessions/week using a home-based one-exercise program: a randomized dose-response trial of knee-extensor resistance exercise in patients eligible for knee replacement (the QUADX-1 trial). Osteoarthritis Cartilage. 2022 Jul;30(7):973-986. doi: 10.1016/j.joca.2022.04.001. Epub 2022 Apr 9. PMID 35413476
- [Background] Elsaman AM, Maaty A, Hamed A. Genicular nerve block in rheumatoid arthritis: a randomized clinical trial. Clin Rheumatol. 2021 Nov;40(11):4501-4509. doi: 10.1007/s10067-021-05821-5. Epub 2021 Jul 2. PMID 34213672
- [Background] Gonzalez Sotelo V, Macule F, Minguell J, Berge R, Franco C, Sala-Blanch X. Ultrasound-guided genicular nerve block for pain control after total knee replacement: Preliminary case series and technical note. Rev Esp Anestesiol Reanim. 2017 Dec;64(10):568-576. doi: 10.1016/j.redar.2017.04.001. Epub 2017 May 26. English, Spanish. PMID 28554709
- [Background] Guler T, Yurdakul FG, Onder ME, Erdogan F, Yavuz K, Becenen E, Uckun A, Bodur H. Ultrasound-guided genicular nerve block versus physical therapy for chronic knee osteoarthritis: a prospective randomised study. Rheumatol Int. 2022 Apr;42(4):591-600. doi: 10.1007/s00296-022-05101-8. Epub 2022 Feb 14. PMID 35165769
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Care Res (Hoboken). 2020 Feb;72(2):149-162. doi: 10.1002/acr.24131. Epub 2020 Jan 6. PMID 31908149